CLINICAL TRIAL: NCT06328335
Title: The Effect of Rehabilitation Training on Orthostatic Hypotension in Parkinson's Patients: a Randomized Controlled Trial
Brief Title: The Effect of Rehabilitation Training on Orthostatic Hypotension in Parkinson's Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copka Sonpashan (Other Government)
Responsible Party: Sponsor-Investigator, Copka Sonpashan, The Research Director, Chao Phya Abhaibhubejhr Hospital
Organization: Chao Phya Abhaibhubejhr Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Orthostatic Hypotension
Record Dates: First submitted 2024-03-10; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Orthostatic Hypotension
MeSH Terms: conditions — Hypotension, Orthostatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive rehabilitation training+Rise-bed Training (Experimental): Assigned by the random number table. During the treatment, all patients were provided with comprehensive rehabilitation therapy as follows:
  Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
  Pulmonary function training, including standing training, cough training, and diaphragm muscle training.
  Interventions: Behavioral: Comprehensive rehabilitation training; Behavioral: Rise-bed Training
- Comprehensive rehabilitation training (Active Comparator): Assigned by the random number table. During the treatment, all patients were provided with comprehensive rehabilitation therapy as follows:
  Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
  Pulmonary function training, including standing training, cough training, and diaphragm muscle training.
  Interventions: Behavioral: Comprehensive rehabilitation training

INTERVENTIONS:
Behavioral: Comprehensive rehabilitation training — Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
  Pulmonary function training, including standing training, cough training, and diaphragm muscle training.
Behavioral: Rise-bed Training — gradually elevating the bed (head-up tilt) is one of the common methods to treat orthostatic hypotension. This treatment adjusts the patient's bed angle to gradually raise their body, promoting balanced blood distribution throughout the body and reducing orthostatic hypotension symptoms.
  In head-up tilt treatment, the bed angle is usually gradually increased from a horizontal position, and the specific angle can be determined based on the patient's condition and tolerance. This treatment process is generally monitored and controlled by medical personnel to ensure safety and effectiveness.
  The mechanism of head-up tilt treatment is to increase venous return by changing the body position and increasing the effect of gravity, thereby increasing cardiac preload, output, and blood pressure. This helps to reduce orthostatic hypotension symptoms such as dizziness, lightheadedness, and fatigue.
  Arms: Comprehensive rehabilitation training+Rise-bed Training

SUMMARY:
The goal of this clinical trial is to explore raise-bed training Orthostatic Hypotension in Parkinson's Patients. The main question it aims to answer is:

Can raise-bed training improve Orthostatic Hypotension in Parkinson's Patients. Patients will be randomly allocated into the control group or the experimental group, all under rehabilitation treatment, the experimental group will be given raise-bed training. The study lasts 21 days for each patient. Researchers will compare Orthostatic Hypotension Questionnaire, Orthostatic Grading Scale, Composite Autonomic Symptom Scale 31 to see if raise-bed training can help improve the symptom

DETAILED DESCRIPTION:
Orthostatic Hypotension is common in Parkinson's Patients. The goal of this clinical trial is to explore raise-bed training Orthostatic Hypotension in Parkinson's Patients. The main question it aims to answer is:

Can raise-bed training improve Orthostatic Hypotension in Parkinson's Patients. Patients will be randomly allocated into the control group or the experimental group, all under rehabilitation treatment, the experimental group will be given raise-bed training. The study lasts 21 days for each patient. Researchers will compare Orthostatic Hypotension Questionnaire, Orthostatic Grading Scale, Composite Autonomic Symptom Scale 31 to see if raise-bed training can help improve the symptom.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Parkinson's disease
* Presence of orthostatic hypotension, defined as a decrease in systolic blood pressure of at least 20 mmHg or a decrease in diastolic blood pressure of at least 10 mmHg within three minutes of standing up
* Age 40 years or older
* Willingness to participate in the study and provide informed consent

Exclusion Criteria:

* Severe cardiovascular disease or other medical conditions that would make head-up tilt treatment unsafe or inappropriate
* Use of medications that affect blood pressure or heart rate, such as beta-blockers or vasodilators, and inability or unwillingness to discontinue these medications for the study period
* History of syncope or falls within the past six months
* Inability to stand or sit up independently or tolerate changes in body position
* Cognitive impairment or inability to provide informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Composite Autonomic Symptom Scale 31 | day 1 and day 21
  The scale has a total score range of 0 to 100, with higher scores indicating a higher symptom burden.
  In this case, a higher score suggests a greater presence of autonomic symptoms, including orthostatic hypotension.

SECONDARY OUTCOMES:
Orthostatic Hypotension Questionnaire | day 1 and day 21
  The Orthostatic Hypotension Questionnaire score ranges 0 to 100 Higher scores on the Orthostatic Hypotension Questionnaire indicate more severe symptoms and a greater impact on quality of life.
Orthostatic Grading Scale | day 1 and day 21
  The Orthostatic Grading Scale is typically graded from 0 to 3, with 0 representing no orthostatic hypotension symptoms and 3 representing severe symptoms.
  In this case, a lower score on the Orthostatic Grading Scale indicates less severe orthostatic hypotension.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Study Chair — Site Coordinator of United Medical Group